CLINICAL TRIAL: NCT04964973
Title: Effect of Transcutaneous Electro-stimulation in Ambulatory Postoperative Rehabilitation Treatment in Thoracic Surgery: Randomized Clinical Trial.
Brief Title: Effect of Transcutaneous Electro-stimulation in Ambulatory Postoperative Rehabilitation Treatment in Thoracic Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Daniel David Álamo Arce, Physical Therapy, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIC 15012
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Thoracic; Postoperative Pain
Keywords: Rehabilitation; Transcutaneous Electric Nerve Stimulation; Thoracic surgery; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The principal investigator and the patient do not know which technique will be applied. The principal investigator and the patients do not know which group they are in, intervention, placebo or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): 1. Control group. Patients have performed the conventional postsurgical program without adding TENS.
  Interventions: Device: Control
- Experimental Group (Experimental): Experimental group. The application of TENS has been added to the physiotherapy program. It had a frequency of 100 Hz and a phase duration of 100 µsec for a period of 30 minutes (through channel 1 of the TENS equipment), receiving and feeling the patient the physical sensation of the current.
  Interventions: Device: Experimental
- Placebo Group (Placebo Comparator): Placebo group. In this group, the same program as group 2 was proposed, using, in this case, channel 2, which did not activate the electric current, and the patient did not receive any physical sensation
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Control — Post-surgical physiotherapeutic activity.
  Arms: Control Group
Device: Experimental — Post-surgical physiotherapeutic activity with the application of the technique
  Arms: Experimental Group
Device: Placebo — Post-surgical physiotherapeutic activity with the application of the non-activated technique
  Arms: Placebo Group

SUMMARY:
Chest pain is one of the most difficult problems to solve after thoracic surgery. Its correct control is often quite difficult, which can cause complications due to an ineffective cough and superficial respiratory movements. It could provoke secretion retention, lung atelectasis, and even pneumonia. In addition, insufficient treatment of postoperative pain also causes a slower recovery of mobility, delaying the incorporation to daily life activities.

Transcutaneous electrical stimulation (TENS) is a technique that attempts to establish pain control by applying electrical current through superficial electrodes Is transcutaneous electrical nerve stimulation effective for the pain rehabilitation approach after thoracic surgery? Are there spirometry changes related to pulmonary function after the application of transcutaneous electrical nerve stimulation in postoperative rehabilitation of thoracic surgical patients?

DETAILED DESCRIPTION:
All patients likely to be part of the study will have an exhaustive medical history. Said clinical history will have, as a basis, the following aspects:

* Filiation data.
* Personal history.
* Type of intervention carried out.
* Incisions made.
* Chronology, location and characteristics of pain. Once intervened, the data corresponding to the surgical intervention performed will be collected. Once the period of 7 days after the intervention has passed and in the absence of complications and pleural drainage, the period of respiratory physiotherapy will begin.

Assessment of quality of life The SF-36 (Short Form Health Survey) health questionnaire will be carried out. This questionnaire is used in medical and mental health research and, in general, in health-related research. It offers an overview of the health status of the person, with the advantage that it is quick and easy to fill out, while also being easy to assess. In the same way, by allowing the numerical assessment of different aspects of the health of the person, it becomes an excellent tool for any research related to health. It contains 36 questions that address different aspects related to the daily life of the person who fills in the questionnaire. These questions are grouped and measured in 8 sections that are evaluated independently and give rise to 8 dimensions that the questionnaire measures.

The eight dimensions are:

1. Physical functioning.
2. Limitation due to physical problems.
3. Body pain.
4. Functioning or social role.
5. Mental health.
6. Limitation due to emotional problems.
7. Vitality, energy or fatigue.
8. General perception of health. In 1991, the project known as "International Quality of Life Assessment" (International Quality of Life Assessment Project, IQOLA) was started, which basically consists of adapting and testing the intercultural applicability of a generic instrument called the SF-Health Survey. (Short Form 36 Health Survey).

The Spanish version of the SF-36 is one of the most widely used generic instruments in the national territory, both in descriptive studies that measure the impact on HRQL in different patient populations and for the evaluation of therapeutic interventions.

Pain assessment

The necessary tools to make a correct pain assessment. In this sense, two ways of measuring it will be established:

1. Self-reports, where the visual analog scale (VAS) will be the basic measurement tool. The pain will be marked with a scale from 0 (absence of pain) to 10 (maximum possible pain).
2. The standardized tests, as an objective of the study, are also proposed to analyze sensitive, affective and behavioral aspects of pain in these patients, it is for this reason that the Mc Gill test will be the tool to take into account.

Assessment of respiratory function The different respiratory parameters will be measured by spirometry (Siebel spirometer): Forced Vital Capacity (FVC); Forced expiratory volume of the first second (FEV1); FEV1 / FVC (Tiffeneau Index).

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent.
* Affected by pulmonary or mediastinal pathology.
* Who have required thoracic surgery.

Exclusion Criteria:

* Patients with pacemakers.
* Diseases with chronic need for analgesic drug.
* History of drug addiction.
* Patients who do not require hospital readmission after surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Spirometry | Six month
  It will consist of a simple spirometry using the Datospir Micro Sibelmed spirometer. The values of the forced vital capacity (FVC) and the volume expired forged in the first second (FEV1) are shown in percentages according to the theoretical values
McGill Test | Six month
  A McGill test will be performed to analyze the level of immediate postoperative pain. The McGill test (Painting Classification Index) (PRI) measures three dimensions: sensory, affective, and evaluative. It consists of 66 words (pain descriptors).
Quality of life survey sf-36 | Six month
  The SF-36 Questionnaire is one of the most used and evaluated Health-Related Quality of Life (HRQOL) instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel David Álamo Arce, P.T., Principal Investigator — Teaching professor and researcher
Locations (1):
- University Hospital of Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wenk M, Schug SA. Perioperative pain management after thoracotomy. Curr Opin Anaesthesiol. 2011 Feb;24(1):8-12. doi: 10.1097/ACO.0b013e3283414175. PMID 21084984
- [Background] Husch HH, Watte G, Zanon M, Pacini GS, Birriel D, Carvalho PL, Kessler A, Sbruzzi G. Effects of Transcutaneous Electrical Nerve Stimulation on Pain, Pulmonary Function, and Respiratory Muscle Strength After Posterolateral Thoracotomy: A Randomized Controlled Trial. Lung. 2020 Apr;198(2):345-353. doi: 10.1007/s00408-020-00335-4. Epub 2020 Feb 8. PMID 32036406
- [Background] Fiorelli A, Morgillo F, Milione R, Pace MC, Passavanti MB, Laperuta P, Aurilio C, Santini M. Control of post-thoracotomy pain by transcutaneous electrical nerve stimulation: effect on serum cytokine levels, visual analogue scale, pulmonary function and medication. Eur J Cardiothorac Surg. 2012 Apr;41(4):861-8; discussion 868. doi: 10.1093/ejcts/ezr108. Epub 2011 Dec 16. PMID 22219414
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Solak O, Turna A, Pekcolaklar A, Metin M, Sayar A, Solak O, Gurses A. Transcutaneous electric nerve stimulation for the treatment of postthoracotomy pain: a randomized prospective study. Thorac Cardiovasc Surg. 2007 Apr;55(3):182-5. doi: 10.1055/s-2006-924631. PMID 17410506
- [Derived] Alamo-Arce DD, Lopez-Fernandez D, Medina-Ramirez R, Vilchez-Barrera M, Etopa-Bitata P, Del Pino Quintana-Montesdeoca M, Baez-Suarez A, Freixinet JL. Effect of transcutaneous electro-stimulation in postoperative rehabilitation pain treatment in thoracic surgery: a randomized clinical trial. Trials. 2024 Dec 19;25(1):839. doi: 10.1186/s13063-024-08613-9. PMID 39702343

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04964973/Prot_000.pdf
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04964973/ICF_001.pdf